CLINICAL TRIAL: NCT00130065
Title: The Effect of Folic Acid Supplementation on Efficacy of Sulfadoxine-pyrimethamine in Pregnant Women in Western Kenya
Brief Title: The Effect of Folic Acid on Efficacy of Sulfadoxine-pyrimethamine in Pregnant Women in Western Kenya
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other); Kenya Ministry of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDC-NCID-3683; UR6-CCU018970
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Malaria
Keywords: Malaria; Pregnancy; Sulfadoxine-pyrimethamine; Folic acid; Folate
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Folic Acid

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine/folic acid
Drug: Sulfadoxine-pyrimethamine/placebo

SUMMARY:
The purpose of this study is to determine whether folic acid, which is often routinely given to pregnant women to prevent birth defects and anemia, affects the efficacy of sulfadoxine-pyrimethamine, another drug that is routinely given to pregnant women in highly malarious areas, for prevention of the adverse effects of malaria during pregnancy.

DETAILED DESCRIPTION:
In malaria endemic areas in sub-Saharan Africa, pregnant women, especially primi- and secundi-gravidae, are more likely to have placental and peripheral parasitemia with Plasmodium falciparum than non-pregnant women. Adverse consequences of malaria in pregnancy include maternal anemia, and low birth weight of the new born. Low birth weight is known to be the most important risk factor for infant mortality.

Intermittent preventive treatment (IPT) with sulfadoxine-pyrimethamine (SP) during pregnancy can mitigate the adverse effects of malaria in pregnancy and is the current standard of care in areas of high malaria transmission in sub-Saharan Africa, as recommended by the World Health Organization.

SP acts by inhibiting parasite enzymes in the metabolism of folic acid. However, in vitro studies indicate that folic acid can antagonize the antimalarial parasite activity of SP. Furthermore, in one West African study, supplementary folic acid compromised the antimalarial efficacy of SP in children with acute malaria aged 6 months to 12 years.

Folic acid requirements are increased during pregnancy, and supplementation with folic acid in pregnancy is recommended. Although in most countries a daily supplementation of 400 to 600 micrograms is considered sufficient, for logistical reasons the daily recommended dose in Kenya is 5 mg of folic acid during pregnancy. It is unknown whether folic acid supplementation might compromise the efficacy of IPT with SP in pregnant women living in malaria endemic areas.

Several studies have shown that HIV-seropositive pregnant women have a higher risk of malaria than HIV-seronegative pregnant women. In addition, HIV-infected women are more likely to be anemic compared with HIV-uninfected women. A few studies have also shown that HIV-seropositive women do not appear to respond as well to IPT with SP compared to HIV-seronegative pregnant women.

In a recent study in pregnant women in Zimbabwe, HIV-infection was a negative predictor of serum folate, and the authors suggested this may be because of reduced intake and absorption, and increased catabolism in HIV-infected pregnant women. Because HIV-seropositive women as a group may have a different folic acid status (and a potential different reaction to folic acid supplementation) than HIV-seronegative women, it is important to assess HIV-status in study participants. It is also important to confirm that no difference exists between HIV-seropositive and HIV-seronegative women in efficacy of SP for clearance of peripheral parasitemia.

Comparison: Parasitemic pregnant women are randomized to receive either SP with folic acid 5 mg, or SP with folic acid 0.4 mg, or SP and placebo. The placebo and the folic acid 0.4 mg are given for two weeks, and then are replaced by folic acid 5 mg.

ELIGIBILITY:
Inclusion Criteria:

* Parasitemia with a parasite density of ≥ 500 parasites/microliter
* Gestational age > 16 weeks and < 35 weeks
* Willingness to provide blood samples and participate in HIV counseling and testing
* Available for follow up for the entire study period
* Hemoglobin > 7 g/dl
* Age 15-45 years

Exclusion Criteria:

* Use of folate in the last 4 weeks
* Gestational age <16 weeks or >35 weeks
* History of an allergy to sulfonamides or other unknown drugs
* Intake of sulfa-containing drugs or 4-aminoquinolones in the previous month
* A urine test positive for sulfa-compounds
* Sickle cell disease
* Concomitant diseases needing treatment with co-trimoxazole or other sulfa-containing drug
* Hemoglobin < 7 g/dl
* Severe malaria or any other serious medical condition requiring hospitalization and/or additional treatment. Clinical danger signs of severe malaria include prostration, impaired consciousness, respiratory distress, multiple convulsions, circulatory collapse, pulmonary oedema, abnormal bleeding, jaundice, and hemoglobinuria. Laboratory signs of severe malaria include severe anemia (hemoglobin < 7 g/dl), hypoglycemia, acidosis, hyperlactataemia, hyperparasitaemia (a parasitemia > 100,000 parasites/µl), and renal impairment

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600
Dates: Start 2003-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Peripheral parasitemia
Hemoglobin level

SECONDARY OUTCOMES:
Effect of HIV serostatus on drug efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Annemieke Van Eijk, M.D., Ph.D., Principal Investigator — Centers for Disease Control and Prevention, Kenya Medical Research Institiute; Monica Parise, M.D., Principal Investigator — Centers for Disease Control and Prevention; Laurence Slutsker, M.D., Principal Investigator — Centers for Disease Control and Prevention, Kenya Medical Research Institute
Locations (1):
- CDC/Kenya Medical Research Institute, Kisumu, Kenya

REFERENCES:
- [Derived] van Eijk AM, Ouma PO, Williamson J, Ter Kuile FO, Parise M, Otieno K, Hamel MJ, Ayisi JG, Kariuki S, Kager PA, Slutsker L. Plasma folate level and high-dose folate supplementation predict sulfadoxine-pyrimethamine treatment failure in pregnant women in Western kenya who have uncomplicated malaria. J Infect Dis. 2008 Nov 15;198(10):1550-3. doi: 10.1086/592715. PMID 18831691